CLINICAL TRIAL: NCT04400487
Title: A Phase 4, Multicenter, Open-label Study to Evaluate the Treatment Effect of Voxelotor on Physical Activity in Adolescents and Adults With Sickle Cell Disease
Brief Title: Actigraphy Improvement With Voxelotor (ActIVe) Study
Acronym: ActIVe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-039; C5341024 (Other: Alias Study Number)
Record Dates: First submitted 2020-03-25; First posted 2020-05-22 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Voxelotor (Experimental): Participants will receive voxelotor at 1500 mg
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — 500 mg Tablet, Oral, With or Without Food
  Other Names: GBT440; Oxbryta

SUMMARY:
This is a study to evaluate the effect of voxelotor on daily physical activity and sleep quality, as measured by a wrist-worn device in participants with sickle cell disease (SCD) and chronic moderate anemia.

DETAILED DESCRIPTION:
All participants will receive Voxelotor as treatment. There will be approximately 13 sites in the US.

Participant safety and tolerability will be monitored during the study using standard measures, including physical examinations, vital signs (including temperature, blood pressure, pulse rate, respiratory rate and peripheral oxygen saturation [SpO2]), clinical laboratory tests, and adverse event (AE) monitoring.

Screening Period (up to 4 weeks in duration): During this period, participants will sign the informed consent form (ICF), after which they will complete the screening assessments as detailed in the Schedule of Assessments (SOA).

Run-in Period (2 weeks in duration): During this period, participants will enter a 2-week run-in period (Day -14 to Day -1) during which baseline actigraphy measures of physical activity and sleep quality, overnight pulse oximetry assessments of oxygen saturation, and Patient-Reported Outcome (PRO) assessments will be collected before initiating treatment with voxelotor.

Treatment Period (24 weeks in duration): After completion of the 14-day Run-in Period, participants will enter the open label treatment period and receive voxelotor 1500 mg once daily for 24 weeks. Repeat actigraphy assessments of physical activity and sleep quality, and overnight pulse oximetry will be performed during the treatment period (Weeks 10 to 12 and Weeks 22 to 24). PRO and Clinical Global Impression (CGI) assessments will be completed at scheduled study visits. The open-label treatment period is considered the continuous 24 weeks of voxelotor treatment from date of first dose (Day 1).

Follow-up Period (4 weeks in duration): Immediately following the 24-week treatment period, participants will enter a 4-week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with SCA (sickle hemoglobin with two sickle cell genes [HbSS] or sickle hemoglobin (S) and one beta thalassemia gene [HbS β0] thal genotype)
2. Between 12 to 55 years of age (inclusive)
3. Screening Hb level ≤8.0 g/dL
4. Treatment with hydroxyurea (HU) therapy on study is permitted if the participant has been on a stable dose for at least 90 days before enrollment with no dose modifications planned or anticipated by the Investigator
5. Treatment with glutamine is permitted
6. Treatment with erythropoiesis-stimulating agents (ESAs) is permitted if the participant has been on a stable dose for at least 12 weeks before enrollment with no dose modifications planned or anticipated by the Investigator
7. Female participants of child-bearing potential must use highly effective methods of contraception to 30 days after the last dose of study drug. Male participants must use barrier methods of contraception to 30 days after the last dose of study drug
8. Females of child-bearing potential are required to have a negative pregnancy test before the administration of study drug
9. Written informed consent and/or parental/guardian consent and participant assent per Institutional Review Board (IRB) policy and requirements, consistent with ICH guidelines

Exclusion Criteria:

1. Red blood cell (RBC transfusion within 3 months before initiation of study drug
2. Planned initiation of regularly scheduled RBC transfusion therapy (also termed chronic, prophylactic, or preventive transfusion) during the study
3. Hospitalization for vaso-occlusive crisis (VOC) or acute chest syndrome (ACS) within 30 days prior to informed consent/assent.
4. More than 10 VOCs requiring hospitalization, emergency department or clinic visit within the past 12 months
5. Planned elective surgery within the next 6 months
6. Physical inactivity attributable to clinically significant musculoskeletal, cardiovascular, or respiratory comorbidities
7. Anemia due to bone marrow failure (eg, myelodysplasia)
8. Absolute reticulocyte count (ARC) < 100 x10^9/L
9. Screening alanine aminotransferase (ALT) > 4× upper limit of normal (ULN)
10. Severe renal dysfunction (estimated glomerular filtration rate [GFR] < 30 mL/min/1.73 m2 by Schwartz formula) or is on chronic dialysis
11. Known active hepatitis A, B or C or known to be human immunodeficiency virus (HIV)-positive.
12. Females who are breast-feeding or pregnant
13. Major surgery within 8 weeks before enrollment. Participants must have completely recovered from any previous surgery before enrollment
14. History of hematopoietic stem cell transplant or gene therapy
15. Received an investigational drug within 30 days or 5-half-lives, whichever is longer, prior to consent, or is currently participating in another trial of an investigational or marketed drug (or medical device)
16. Use of concomitant medications (eg, crizanlizumab) that confound the ability to interpret data from the study
17. Medical, psychological, or behavioral condition that, in the opinion of the Investigator, would confound or interfere with evaluation of safety and/or efficacy of the study drug, prevent compliance with the study protocol; preclude informed consent; or, render the participant unable/unlikely to comply with the study procedures
18. Use of herbal medications (e.g., St. John's Wort), sensitive cytochrome P450 (CYP) 3A4 substrates with a narrow therapeutic index, strong CYP3A4 inhibitors, fluconazole, or moderate or strong CYP3A4 inducers
19. Symptomatic coronavirus disease of 2019 (COVID-19) infection

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - UConn Health, Farmington, Connecticut
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Hospital of Michigan, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Duke Department of Pediatrics, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - VCU Health, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a 28-day screening period, a 14-day run-in period, a 24-week treatment period and a 28-day follow-up period after last dose.
Pre-assignment Details: A total of 25 participants were enrolled in the study.
Groups:
- Voxelotor: Participants received 1500 milligram (mg) of voxelotor (three tablets of 500 mg) orally once daily for 24 weeks (168 days).
Period: Screening Period (28 Days)
Arm/Group | Voxelotor
Started | 25
Completed | 25
Not Completed | 0
Period: Run-in Period (14 Days)
Arm/Group | Voxelotor
Started | 25
Completed | 25
Not Completed | 0
Period: Treatment Period (24 Weeks)
Arm/Group | Voxelotor
Started | 25
Treated (With at Least 1 Dose of Study Treatment) | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance | 1
Period: Follow-up Period (28 Days)
Arm/Group | Voxelotor
Started | 23
Completed | 21
Not Completed | 2
Not completed — Started commercial product | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study treatment were included in the safety population.
Arm/Group | Voxelotor
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Daily Physical Activity (Counts Per Minute) to Week 10-12
Description: Daily physical activity was measured by actigraphy in participants with sickle cell disease (SCD) and chronic moderate anemia. Actigraphy assessments were performed using wrist-worn tri-axial accelerometry device. Actigraphy is an accepted methodology for tracking activity levels, time spent in moderate and vigorous physical activity, step counts, and energy expenditure. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments. In this outcome measure the average of at least 8 valid days during the specified two-week period was considered. A participant's daily wear must be 18 hours or more in a day to be considered a valid day.
Time Frame: Baseline, Week 10-12
Population: Participants who received at least 1 dose of voxelotor were included in the safety population. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Counts per minute
Arm/Group | Voxelotor
Number analyzed (Participants) | 16
Counts per minute | -155.6 (458.45)

2. Primary Outcome: Change From Baseline in Total Daily Physical Activity (Counts Per Minute) to Week 22-24
Description: Daily physical activity was measured by actigraphy in participants with SCD and chronic moderate anemia. Actigraphy assessments were performed using wrist-worn tri-axial accelerometry device. Actigraphy is an accepted methodology for tracking activity levels, time spent in moderate and vigorous physical activity, step counts, and energy expenditure. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments. In this outcome measure the average of at least 8 valid days during the specified two-week period was considered. A participant's daily wear must be 18 hours or more in a day to be considered a valid day.
Time Frame: Baseline, Week 22-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Counts per minute
Arm/Group | Voxelotor
Number analyzed (Participants) | 14
Counts per minute | -79.4 (443.77)

3. Primary Outcome: Change From Baseline in Light Physical Activity to Week 10-12
Description: Change in daily physical activity was measured by actigraphy in adolescent and adult participants with SCD and chronic moderate anemia. This outcome measure described the change from baseline in light physical activity. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments. In this outcome measure the average of at least 8 valid days during the specified two-week period was considered. A participant's daily wear must be 18 hours or more in a day to be considered a valid day.
Time Frame: Baseline, Week 10-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 16
minutes/day | 5.8 (62.67)

4. Primary Outcome: Change From Baseline in Light Physical Activity to Week 22-24
Description: as for outcome 3
Time Frame: Baseline, Week 22-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 14
minutes/day | -11.7 (115.34)

5. Primary Outcome: Change From Baseline in Moderate Physical Activity to Week 10-12
Description: Change in daily moderate physical activity (minutes per day) was measured by actigraphy in participants with SCD and chronic moderate anemia. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments. In this outcome measure the average of at least 8 valid days during the specified two-week period was considered. A participant's daily wear must be 18 hours or more in a day to be considered a valid day.
Time Frame: Baseline, Week 10-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 16
minutes/day | -9.0 (25.55)

6. Primary Outcome: Change From Baseline in Moderate Physical Activity to Week 22-24
Description: as for outcome 5
Time Frame: Baseline, Week 22-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 14
minutes/day | -5.7 (30.01)

7. Primary Outcome: Change From Baseline in Vigorous Physical Activity to Week 10-12
Description: Change in daily vigorous physical activity (minutes per day) was measured by actigraphy in participants with SCD and chronic moderate anemia. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments. In this outcome measure the average of at least 8 valid days during the specified two-week period was considered. A participant's daily wear must be 18 hours or more in a day to be considered a valid day.
Time Frame: Baseline, Week 10-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 16
minutes/day | 0.0 (4.94)

8. Primary Outcome: Change From Baseline in Vigorous Physical Activity to Week 22-24
Description: as for outcome 7
Time Frame: Baseline, Week 22-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 14
Minutes/day | -1.2 (6.52)

9. Primary Outcome: Change From Baseline in Total Nocturnal Sleep Time to Week 10-12
Description: Total nocturnal sleep time was measured by overnight actigraphy monitoring. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments. In this outcome measure the average of at least 8 valid days during the specified two-week period was considered. A participant's daily wear must be 18 hours or more in a day to be considered a valid day.
Time Frame: Baseline, Week 10-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 16
Minutes/day | 0.3 (77.64)

10. Primary Outcome: Change From Baseline in Total Nocturnal Sleep Time to Week 22-24
Description: as for outcome 9
Time Frame: Baseline, Week 22-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 14
Minutes/day | 17.6 (141.10)

11. Primary Outcome: Change From Baseline in Wake Time After Sleep Onset to Week 10-12
Description: Measured by actigraphy monitoring. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments. In this outcome measure the average of at least 8 valid days during the specified two-week period was considered. A participant's daily wear must be 18 hours or more in a day to be considered a valid day.
Time Frame: Baseline, Week 10-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 16
Minutes/day | 2.0 (37.10)

12. Primary Outcome: Change From Baseline in Wake Time After Sleep Onset to Week 22-24
Description: as for outcome 11
Time Frame: Baseline, Week 22-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | Voxelotor
Number analyzed (Participants) | 14
Minutes/day | 2.0 (42.00)

13. Primary Outcome: Change From Baseline in Sleep Efficiency to Week 10-12
Description: Sleep efficiency was defined as ration of total sleep time to time in bed. Change from baseline to follow-up visit was calculated as the baseline measurement subtracted from the follow-up measurement for all assessments.
Time Frame: Baseline, Week 10-12
Population: Data for this outcome measure could not be analyzed and reported as data for 'time in bed' was not collected which was required to calculate sleep efficiency.
Arm/Group | Voxelotor
Number analyzed (Participants) | 0

14. Primary Outcome: Change From Baseline in Sleep Efficiency to Week 22-24
Description: as for outcome 13
Time Frame: Baseline, Week 22-24
Population: as for outcome 13
Arm/Group | Voxelotor
Number analyzed (Participants) | 0

15. Primary Outcome: Percentage of Participants With a More Than (>)1 Grams Per Deciliter (g/dL) Increase in Hemoglobin (Hb) at Week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Voxelotor
Number analyzed (Participants) | 24
Percentage of participants | 41.7

16. Primary Outcome: Percentage of Participants With a >1 g/dL Increase in Hemoglobin (Hb) at Week 24
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Voxelotor
Number analyzed (Participants) | 23
Percentage of participants | 26.1

17. Primary Outcome: Change From Baseline in Mean Overnight Oxygen Saturation (SpO2 Percentage [%]) to Week 10-12
Time Frame: Baseline, Week 10-12
Population: Data for this outcome measure was not analyzed and reported because SpO2 data was not collected as the device that was supposed to measure SpO2 did not work.
Arm/Group | Voxelotor
Number analyzed (Participants) | 0

18. Primary Outcome: Change From Baseline in Mean Overnight SpO2 % to Week 22-24
Time Frame: Baseline, Week 22-24
Population: as for outcome 17
Arm/Group | Voxelotor
Number analyzed (Participants) | 0

19. Primary Outcome: Change From Baseline in Median Number of Overnight SpO2 Dips > 3% Per Hour to Week 10-12
Time Frame: Baseline, Week 10-12
Population: as for outcome 17
Arm/Group | Voxelotor
Number analyzed (Participants) | 0

20. Primary Outcome: Change From Baseline in Median Number of Overnight SpO2 Dips > 3% Per Hour to Week 22-24
Time Frame: Baseline, Week 22-24
Population: as for outcome 17
Arm/Group | Voxelotor
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From screening period to 28 days post last dose of study treatment (maximum of 238 days)
Description: All participants who received at least 1 dose of study treatment were included in the safety population. Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other, or a participant may have experienced both serious and non-serious event. AEs were presented which were related to both SCD and Non-SCD related.
Groups:
- Voxelotor: SCD Related: Participants who received voxelotor 1500 mg and had SCD related AEs.
- Voxelotor: Non-SCD Related: Participants received voxelotor 1500 mg and had non-SCD related AEs.
Arm/Group | Voxelotor: SCD Related | Voxelotor: Non-SCD Related
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 8/25 | 3/25
Other Adverse Events (participants affected / at risk) | 5/25 | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voxelotor: SCD Related (N=25) | Voxelotor: Non-SCD Related (N=25)
Cellulitis (Infections and infestations) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 8 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voxelotor: SCD Related (N=25) | Voxelotor: Non-SCD Related (N=25)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 9
Nausea (Gastrointestinal disorders) | 0 | 6
Vomiting (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 6
Dizziness (Nervous system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2
Scrotal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT04400487/Prot_000.pdf